CLINICAL TRIAL: NCT05155124
Title: Safety of Cetuximab in Combination With Trifluridin Tipiracil in the Third-line Treatment of RASwt Metastatic Colorectal Cancer
Brief Title: Safety of Cetuximab and Trifluridin Tipiracil as the Third-line Therapy in the RASwt mCRC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hongli Liu, Director, Head of GI Department , Principal Investigator, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT001
Record Dates: First submitted 2021-12-07; First posted 2021-12-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Neoplasms Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab and trifluridin tipiracil (Experimental): Cetuximab will be administered at a fixed dose of 500 mg/m2 once every 2 weeks; trifluridin tipiracil will be administered in a dose de-escalation design: dose level 1: 35 mg/m2 twice daily on days 1-5 once every 2 weeks; Or dose level 0: 30 mg/m2, twice daily, Days 1-5, once every 2 weeks;
  Interventions: Drug: Cetuximab + trifluridin tipiracil

INTERVENTIONS:
Drug: Cetuximab + trifluridin tipiracil — Cetuximab will be administered at a fixed dose of 500 mg/m2 once every 2 weeks; trifluridin tipiracil will be administered in a dose de-escalation design: dose level 1: 35 mg/m2 twice daily on days 1-5 once every 2 weeks; Or dose level 0: 30 mg/m2, twice daily, Days 1-5, once every 2 weeks;
  Other Names: Erbitux；TAS102;TAS-102

SUMMARY:
This was a single-arm, prospective study to investigate the safety of cetuximab in combination with trifluridin tipiracil (TAS-102) in the third-line treatment of Chinese patients with RAS wild-type mCRC.

DETAILED DESCRIPTION:
This was a single-arm, prospective study to investigate the safety of cetuximab in combination with trifluridin tipiracil (TAS-102) in the third-line treatment of Chinese patients with RAS wild-type mCRC. Cetuximab will be administered at a fixed dose of 500 mg/m2 once every 2 weeks; trifluridin tipiracil will be administered in a dose de-escalation design: dose level 1: 35 mg/m2 twice daily on days 1-5 once every 2 weeks; after 1 cycle will be observed, and if ≤ 2 patients experience DLT, this dose level will be the recommended phase II dose; if ≥ 3 patients experience DLT, additional 6 patients will receive dose level 0. ( Dose level 0: 30 mg/m2, twice daily, Days 1-5, once every 2 weeks;) If ≤ 2 individuals experience DLT, this dose level is the recommended Phase II dose; if ≥ 3 individuals experience DLT, the study will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old male or female;
* Histologically or cytologically confirmed metastatic colon or rectal adenocarcinoma; excluding appendiceal cancer and anal canal cancer;
* Previously received second-line treatment, at least 2 standard chemotherapy regimens(including fluorouracil, capecitabine, irinotecan, oxaliplatin, raltitrexed and anti-VEGF, anti-EGFR, etc.), if already accepted anti-EGFR treatment achieved at least PR or above;
* ECOG PS 0-1;
* At least one measurable lesion by CT or MRI (according to RECIST 1.1 criteria, the longest diameter of tumor lesion CT/MRI scan ≥ 10 mm, lymph node lesion CT/MRI scan shortest diameter ≥ 15 mm);
* RAS gene mutation detection results are wild-type. The test sample can be the primary tumor or metastasis sample;
* Can receive oral drug treatment;
* Normal function of major organs, meeting the following criteria within 14 days before the start of treatment:

  1. neutrophil count ≥ 1.5 × 10*9/L;
  2. Platelet count ≥ 75 × 10*9/L;
  3. Hemoglobin ≥ 9.0 g/dL;
  4. AST ≤ 2.5 × UNL (upper limit of normal) (if liver metastasis AST ≤ 5 × UNL);
  5. ALT ≤ 2.5 × UNL (if liver metastasis AST ≤ 5 × UNL);

  g.Creatinine clearance (calculated according to Cockcroft and Gault formula) > 60 mL/min or serum creatinine ≤ 1.5 × UNL;
* Expected survival time > 3 months (90 days);
* Women of childbearing potential must have used reliable contraception and had a negative pregnancy test within 7 days prior to enrollment and be willing to use an appropriate method of contraception during the trial and for 6 months after the last dose of trial drug. Males must agree to use an adequate method of contraception or have been surgically sterilized during the trial and for 6 months after the last dose of trial drug;
* The patients voluntarily participated in this study and signed the informed consent form, with good compliance and cooperation in the follow-up.

Exclusion Criteria:

* Previously treated with regorafenib, fruquintinib, TAS-102;
* Participated in another drug clinical trial in the past 4 weeks, or received systemic chemotherapy, radiotherapy or biological therapy in the past 4 weeks;
* Known brain metastases or strongly suspected brain metastases;
* Patients with known BARF mutations should be excluded;
* Synchronous cancer or metachronous cancer with disease-free survival ≥ 5 years (except colorectal cancer), excluding mucosal cancer (esophageal cancer, gastric cancer, cervical cancer, non-melanoma skin cancer, bladder cancer, etc.) that has been cured or may be cured by local resection;
* Factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and gastric intestinal obstruction; ucontrolled Crohn's disease or ulcerative colitis;
* Serosal effusion (including pleural effusion, ascites, pericardial effusion) with clinical symptoms and requiring symptomatic treatment;
* Pregnant or lactating women; patients of childbearing potential are unwilling or unable to take effective contraceptive measures;
* Known to be allergic to the study drug, study drug class and its ingredients;
* Conditions requiring systemic steroid treatment (except topical steroid and cetuximab pretreatment);
* History of interstitial lung disease (interstitial pneumonia, pulmonary fibrosis, etc.) or CT findings of interstitial lung disease;
* Active local or systemic infection requiring treatment;
* Cardiac function classification (NYHA classification) ≥ Grade III or severe heart disease;
* Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) or active hepatitis B, C;
* Toxicity not recovered (CTCAE > grade 1) or not completely recovered from previous anticancer surgery;
* Patients judged by the Investigator as unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT（Dose-limited toxicity） | From Baseline to primary completion date, about 18 months
  Determination of RP2D based on incidence of DLT

SECONDARY OUTCOMES:
Adverse Eevents | From Baseline to primary completion date, about 18 months
  Participants With Incidence of Adverse Eevents During Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Liu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No